CLINICAL TRIAL: NCT04041349
Title: Clinical Observation for the Therapeutic Effect of mNGF on Cognitive Decline in Cerebral Small Vessel Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First Affiliated Hospital of Jinan University (Other); Guangdong 999 Brain Hospital (Other); Dongguan People's Hospital (Other Government); Houjie Hospital of Dongguan City (Unknown); First Affiliated Hospital of Shantou University Medical College (Other); Wuhan University (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Responsible Party: Principal Investigator, Gao Xiaoya, Associate Chief Physician, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-KY-026-02
Record Dates: First submitted 2019-07-09; First posted 2019-08-01 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: Cerebral Small Vessel Diseases; Mouse Nerve Growth Factor; cognitive impairment
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The standard treatment group (No Intervention): The standard treatment group is treated with conventional drugs and cholinesterase inhibitors
- mouse nerve growth factor (mNGF)group (Experimental): Conventional drugs and cholinesterase inhibitors + mouse nerve growth factor (mNGF) of 20 μg (9000 U)/day for 14 consecutive days by intramuscular injection.
  Interventions: Drug: mouse nerve growth factor

INTERVENTIONS:
Drug: mouse nerve growth factor — mouse nerve growth factor of 20 UG (9000 U)/day for 14 consecutive days by intramuscular injection
  Other Names: mNGF
  Arms: mouse nerve growth factor (mNGF)group

SUMMARY:
This study was a multicenter, prospective, randomized controlled trial. In this study, 510 patients with cognitive impairment of cerebral small vessel disease who met the inclusion criteria are randomly included in multiple centers and randomized into two groups (standard treatment group and mouse nerve growth factor addition treatment group). The standard treatment group is treated with conventional drugs and cholinesterase inhibitors. In addition to the above treatment, the mouse nerve growth factor addition treatment group is administered with nerve growth factor 20 μg (9000 U)/vial for 14 consecutive days, intramuscularly once a day. Systematic clinical evaluation of patient cognitive function is performed at baseline, 14-day, and 3-month follow-up, and imaging (MR) is also evaluated twice at baseline, 14-day, and 3-month follow-up. At last observe the clinical effect of mouse nerve growth factor on cognitive impairment of cerebral small vessel disease.

DETAILED DESCRIPTION:
Cerebral small vessel disease (CSVD) refers to the disease that involves cerebral small blood vessels, including arterioles, arterioles, capillaries, and venules, etc.The clinical manifestations of CSVD are complex and varied, but cognitive impairment is one of the core clinical manifestations of CSVD, and some patients have gait and sphincter dysfunction.At present, CSVD is an important subtype of vascular cognitive dysfunction and the most common cause of vascular dementia in clinic.Currently, the treatment of cognitive impairment in small cerebral vascular diseases is conducted in two aspects: the treatment and prevention of the structure and function of small cerebral vascular diseases, and the treatment of cognitive dysfunction.The treatments recommended by experts for cognitive dysfunction include cholinesterase inhibitors, nmda-receptor antagonists, and other drugs, but these drugs have not been specifically studied for the treatment of cognitive impairment in small cerebral vascular diseases.The treatment of cognitive impairment in small cerebral vascular disease is still in difficulty, and there is no effective and specific treatment at present.Mouse Nerve Growth Factor (mNGF) is a soluble protein which promotes Nerve Growth, isolated and purified successively by Levi-Montalcini and Cohen in 1959 and 1960.The discovery of NGF makes people realize that some factors are needed to promote the development, growth and maintain the activity of neurons in the process of nervous system, which opens up a new field of neurobiology, for which the two scholars won the 1986 Nobel Prize in physiology.Clinical use of NGF in the treatment of Alzheimer's Disease (AD), NGF injection into Meynert basal ganglia showed that NGF can improve the symptoms of AD and AD induced brain atrophy.Meynert basal ganglia is considered to be the main source of cholinergic neurons and plays an important role in the pathogenesis of AD and Parkinson's Disease (PD). Similar studies in China have also confirmed that nerve growth factor can reduce the symptoms of vascular dementia in stroke patients and delay the development of cognitive dysfunction.It has been found that nerve growth factor, like other special types of macromolecular proteins, can pass through the blood-brain barrier (BBB) through receptor-mediated endocytosis.In the animal studies, BBB integrity was significantly damaged in rats with hypertensive white matter lesions, in which case, nerve growth factor can play a role in protecting neurons, preventing cell apoptosis and promoting nerve reconstruction through BBB.By carrying out this study, the researchers intend to explore the therapeutic effect of rat nerve growth factor on cognitive dysfunction caused by cerebral small vascular disease, and preliminarily explore its imaging mechanism, so as to provide a new direction for further research on drug treatment of cognitive dysfunction caused by cerebral small vascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50-80 years old;
2. Clinical symptoms of acute CSVD, including Transient ischemic attack (TIA) or lacunar infarction, and with related lesions on MRI imaging (acute infarction with diameter < 20mm on (diffusion weighted imaging) DWI or with diameter of 3-15mm on MRI-T1,T2 or FLAIR);
3. For patients with chronic CSVD symptoms, two or more CSVD imaging markers are required : lacune (number > = 1), white matter lesion (Fazekas > = 2), cerebral microbleeds (number > =1 in deep white matter), enlarged perivascular space(number > = 10 in basal ganglia);
4. Clinical diagnosis of vascular cognitive impairment or dementia, MMSE score =<26;
5. Signed informed consent.

Exclusion Criteria:

1. Intracranial or extracranial arterial stenosis of > 50% luminal stenosis or prior history of endarterectomy of cerebral large arteries;
2. TOAST classification suggested (very) possible cardioembolic stroke;
3. Large cortical or subcortical infarction with diameter > 1.5cm on MRI; White matter lesions caused by other diseases such as multiple sclerosis; Other central nervous system diseases such as cerebral hemorrhage, brain trauma, epilepsy, encephalitis, hydrocephalus or brain tumors; Oher systemic diseases, such as liver and kidney insufficiency, tumor, etc.;
4. History of alcohol intoxication, drug addiction, or mental disease, or severe aphasia;
5. Contraindication for MRI examination. -

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-07 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
change of Alzheimer's disease assessment scale-cognition (ADAS-cog) score | Baseline -14 days -3 months
  Cognitive function assessment

SECONDARY OUTCOMES:
change of Mini-mental State Examination (MMSE) | Baseline -14 days -3 months
  Dementia screening scale
Montreal Cognitive Assessment (MoCA) scale | Baseline -14 days -3 months
  A rapid screening tool for mild cognitive impairment
digit span test | Baseline -14 days -3 months
  test the ability to concentrate attention, instantaneous memory and anti - information interference ability
Activity of Daily Living Scale | Baseline -14 days -3 months
  Barthel index was used to reflect the daily life ability of the interviewees
Patient Health Questionnaire-9 Score | Baseline -14 days -3 months
  Depression assessment tool
Hamilton anxiety scale | Baseline -14 days -3 months
  Assess the severity of anxiety symptoms in neurosis and other patients
Hamilton depression scale | Baseline -14 days -3 months
  A commonly used scale in clinical evaluation of depression

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoya Gao, Doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospiatal, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No